CLINICAL TRIAL: NCT06108388
Title: Functional Investigation of Endothelial Function and Regenerative Cell Exhaustion in Type 2 Diabetes
Brief Title: Functional Investigation of Endothelial Function and Regenerative Cell Exhaustion
Acronym: FIERCE
Status: Not yet recruiting | Type: Observational
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: Unity Health Toronto (Other); University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00074548
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes; Vascular regeneration; Hematopoietic progenitor cells; Functionality; EndoPAT; Endothelial dysfunction; scRNA-seq; Colony formation assay; Secretome analyses
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum samples will be retained for 5 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 Diabetes: Participants living with type 2 diabetes for less than 10 years will be recruited.
- No Diabetes: Participants not living with diabetes will be recruited.

SUMMARY:
FIERCE is an observational cross-sectional study. Approximately 90 individuals living with type 2 diabetes (T2D) and/or individuals living without diabetes will be randomized (2:1).

The primary objective of this trial is to determine if there are differences in the content and function of circulating vascular regenerative (VR) progenitor cell subsets isolated from individuals living with T2D versus individuals not living with T2D. The main question this study aims to answer is: Does T2D compromise or enhance VR cell functionality?

Each participant will be asked to provide a single blood sample. Blood samples will be processed to enumerate the number of vessel-repairing cells and determine the functionality of the different subtypes of vessel-repairing cells.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a significant and prevalent global health concern. Individuals diagnosed with T2D are at an elevated risk of developing atherosclerotic cardiovascular (CV) disease, a leading cause of global morbidity and mortality.

Blood vessel homeostasis plays a central role in the status of CV health. Circulating vascular regenerative (VR) progenitor cells, which mediate the endogenous processes of angiogenesis, vasculogenesis, and arteriogenesis, are critical in orchestrating vessel repair. In T2D, chronic hyperglycemia and concomitant oxidative stress create a maladaptive environment that impairs vessel repair. T2D can lead to a chronic state known as vascular regenerative cell exhaustion (VRCE), characterized by the depletion of, and dysfunction in, circulating VR progenitor cells. The available data indicate that VRCE associated with T2D can lead to VR cell dysfunction and compromised vascular repair.

The investigators have developed a multi-parametric flow cytometry assay to measure VR progenitor cell content in blood samples. This assay utilizes the cytosolic detoxification enzyme aldehyde dehydrogenase (ALDH), which is highly expressed in progenitor cells from hematopoietic, endothelial, and mesenchymal stromal cell lineages. This enzyme protects progenitor cells from oxidative damage that is driven by reactive oxygen species. ALDH activity is reduced by up to 100-fold as progenitor cells differentiate towards more expendable effector cells. As such, the investigators identify cells with high or low ALDH activity in combination with cell surface markers to distinguish progenitor cell subsets (ALDHhi) from more differentiated progeny (ALDHlow). Used in conjunction with 'side scatter' (SSC), a parameter that correlates with the granularity or complexity of a cell, this assay can distinguish between and quantify ALDHhiSSClow hematopoietic/endothelial precursor cells, ALDHhiSSCmid monocytes, and ALDHhiSSChi granulocyte precursors. Previously, bone marrow-derived ALDHhiSSClow cells were shown to co-express the primitive cell markers CD34 and CD133 and exhibit multipotent hematopoietic colony-forming ability in vitro. In the immunodeficient NOD/SCID mouse model of hindlimb ischemia, transplantation of ALDHhiSSClow cells into the ischemic limb led to improved muscle perfusion recovery. The potential of this cell therapy to prevent amputations in individuals with critical limb ischemia has been evaluated in clinical trial settings.

The peripheral blood of individuals living with T2D for >10-years exhibits a depletion of ALDHhiSSClow VR progenitor cells, lower frequencies of ALDHhiSSCmid monocytes with vessel reparative function, and an increased frequency of ALDHhiSSChi inflammatory granulocyte precursors compared to that from individuals not living with T2D. The VRCE phenotype was partially reversed in people living with T2D and established coronary artery disease (CAD) after they had been on the SGLT2 inhibitor empagliflozin for 6 months. Obesity-induced VR cell depletion was also reversed by 3 months post-bariatric surgery. These findings collectively provided a mechanistic link between T2D, obesity, and impaired vessel homeostasis/repair, and also established that VRCE may be therapeutically reversed in a high CV-risk diabetic milieu.

FIERCE will assess VR cell content in individuals living with T2D (<10-years duration) and age- and sex-matched individuals not living with T2D. It will also assess the function of circulating ALDHhi VR cells through: (1) Endothelial peripheral arterial tonometry (EndoPAT) to clinically analyze endothelial function through reactive hyperemic index, (2) multipotent hematopoietic colony formation assays in vitro, (3) single-cell RNA-sequencing (scRNA-seq) that is focused on mRNA expression associated with angiogenesis, and (4) quantitative, label-free secretome analyses to determine changes in pro-angiogenic protein secretion.

The investigators hypothesize that VRCE impairs vascular repair and blood vessel regeneration during T2D and is partly caused by impaired pro-angiogenic properties of VR progenitor cell subsets. Specifically, the investigators postulate that multipotent hematopoietic colony formation, pro-angiogenic cytokine mRNA expression, and pro-angiogenic protein release will be lower in ALDHhi progenitor cell subsets from individuals living with T2D relative to participants not living with T2D. The investigators also predict that individuals living with T2D will exhibit a lower reactive hyperemic index compared to individuals not living with T2D.

Characterization of ALDHhi progenitor VR cell dysfunction in the setting of T2D will generate proof-of-concept to support the potential use of VR cell content as a quantifiable and functional indicator of vascular health.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Willing to provide written informed consent.
* Documented history of T2D
* No documented history of diabetes

Exclusion Criteria:

* Unable or unwilling to provide written informed consent or provide a peripheral blood sample.
* Any life-threatening disease expected to result in death within two years of consent.
* Any malignancy not considered cured (except basal cell carcinoma of the skin). An individual is considered cured if there has been no evidence of cancer recurrence for the five years prior to screening.
* Known severe liver disease.
* White blood cell count ≥15 x 10^9/L.
* Active infectious disease requiring systemic antibiotic or anti-viral agents.
* Known acquired immunodeficiency syndrome such as HIV.
* Treated autoimmune disorders (e.g. T1D and LADA).
* On oral steroid therapy (e.g. prednisone or other corticosteroids) or other immunosuppressive agents (e.g. methotrexate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Individuals will be asked their self-representation of their gender identity.
Study Population: Participants will be identified from primary care clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Hematopoietic colony formation in ALDHhiSSClow regenerative cell subsets | Baseline
  The capacity for total multipotent hematopoietic colony formation in ALDHhiSSClow regenerative cell subsets isolated from individuals living with T2D versus individuals not living with T2D.

SECONDARY OUTCOMES:
Endothelial function | Baseline
  Endothelial peripheral arterial tonometry (EndoPAT) will be utilized to clinically analyze endothelial function through reactive hyperemic index in individuals living with T2D and individuals not living with T2D.
Frequency and absolute number of circulating ALDHhiSSClowCD133+ progenitor cells | Baseline
  The change in the frequency and absolute number of circulating ALDHhiSSClowCD133+ progenitor cells between individuals living with T2D versus age- and sex-matched individuals not living with T2D

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — Unity Health Toronto; David A Hess, PhD, Principal Investigator — Robarts Research Institute, London, Ontario
Locations (1):
- Diagnostic Assessment Centre, Scarborough Village, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rawshani A, Rawshani A, Franzen S, Sattar N, Eliasson B, Svensson AM, Zethelius B, Miftaraj M, McGuire DK, Rosengren A, Gudbjornsdottir S. Risk Factors, Mortality, and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2018 Aug 16;379(7):633-644. doi: 10.1056/NEJMoa1800256. PMID 30110583
- [Background] Haas AV, McDonnell ME. Pathogenesis of Cardiovascular Disease in Diabetes. Endocrinol Metab Clin North Am. 2018 Mar;47(1):51-63. doi: 10.1016/j.ecl.2017.10.010. PMID 29407056
- [Background] Hess DA, Verma S, Bhatt D, Bakbak E, Terenzi DC, Puar P, Cosentino F. Vascular repair and regeneration in cardiometabolic diseases. Eur Heart J. 2022 Feb 10;43(6):450-459. doi: 10.1093/eurheartj/ehab758. PMID 34849704
- [Background] Szmitko PE, Fedak PW, Weisel RD, Stewart DJ, Kutryk MJ, Verma S. Endothelial progenitor cells: new hope for a broken heart. Circulation. 2003 Jun 24;107(24):3093-100. doi: 10.1161/01.CIR.0000074242.66719.4A. No abstract available. PMID 12821589
- [Background] Dimmeler S. Regulation of bone marrow-derived vascular progenitor cell mobilization and maintenance. Arterioscler Thromb Vasc Biol. 2010 Jun;30(6):1088-93. doi: 10.1161/ATVBAHA.109.191668. Epub 2010 May 7. PMID 20453167
- [Background] Fadini GP, Miorin M, Facco M, Bonamico S, Baesso I, Grego F, Menegolo M, de Kreutzenberg SV, Tiengo A, Agostini C, Avogaro A. Circulating endothelial progenitor cells are reduced in peripheral vascular complications of type 2 diabetes mellitus. J Am Coll Cardiol. 2005 May 3;45(9):1449-57. doi: 10.1016/j.jacc.2004.11.067. PMID 15862417
- [Background] Fadini GP, Boscaro E, de Kreutzenberg S, Agostini C, Seeger F, Dimmeler S, Zeiher A, Tiengo A, Avogaro A. Time course and mechanisms of circulating progenitor cell reduction in the natural history of type 2 diabetes. Diabetes Care. 2010 May;33(5):1097-102. doi: 10.2337/dc09-1999. Epub 2010 Feb 11. PMID 20150295
- [Background] Mauch P, Hellman S. Loss of hematopoietic stem cell self-renewal after bone marrow transplantation. Blood. 1989 Aug 1;74(2):872-5. PMID 2665859
- [Background] Bigarella CL, Liang R, Ghaffari S. Stem cells and the impact of ROS signaling. Development. 2014 Nov;141(22):4206-18. doi: 10.1242/dev.107086. PMID 25371358
- [Background] Moore MA. Does stem cell exhaustion result from combining hematopoietic growth factors with chemotherapy? If so, how do we prevent it? Blood. 1992 Jul 1;80(1):3-7. No abstract available. PMID 1377052
- [Background] Mangialardi G, Spinetti G, Reni C, Madeddu P. Reactive oxygen species adversely impacts bone marrow microenvironment in diabetes. Antioxid Redox Signal. 2014 Oct 10;21(11):1620-33. doi: 10.1089/ars.2014.5944. PMID 25089632
- [Background] Terenzi DC, Trac JZ, Teoh H, Gerstein HC, Bhatt DL, Al-Omran M, Verma S, Hess DA. Vascular Regenerative Cell Exhaustion in Diabetes: Translational Opportunities to Mitigate Cardiometabolic Risk. Trends Mol Med. 2019 Jul;25(7):640-655. doi: 10.1016/j.molmed.2019.03.006. Epub 2019 Apr 30. PMID 31053416
- [Background] Hayden J, O'Donnell G, deLaunois I, O'Gorman C. Endothelial Peripheral Arterial Tonometry (Endo-PAT 2000) use in paediatric patients: a systematic review. BMJ Open. 2023 Jan 18;13(1):e062098. doi: 10.1136/bmjopen-2022-062098. PMID 36657756
- [Background] Li Q, Wang M, Zhang S, Jin M, Chen R, Luo Y, Sun X. Single-cell RNA sequencing in atherosclerosis: Mechanism and precision medicine. Front Pharmacol. 2022 Oct 4;13:977490. doi: 10.3389/fphar.2022.977490. eCollection 2022. PMID 36267275
- [Background] Kehl D, Generali M, Mallone A, Heller M, Uldry AC, Cheng P, Gantenbein B, Hoerstrup SP, Weber B. Proteomic analysis of human mesenchymal stromal cell secretomes: a systematic comparison of the angiogenic potential. NPJ Regen Med. 2019 Apr 16;4:8. doi: 10.1038/s41536-019-0070-y. eCollection 2019. PMID 31016031
- [Result] GBD 2021 Diabetes Collaborators. Global, regional, and national burden of diabetes from 1990 to 2021, with projections of prevalence to 2050: a systematic analysis for the Global Burden of Disease Study 2021. Lancet. 2023 Jul 15;402(10397):203-234. doi: 10.1016/S0140-6736(23)01301-6. Epub 2023 Jun 22. PMID 37356446
- [Result] Putman DM, Liu KY, Broughton HC, Bell GI, Hess DA. Umbilical cord blood-derived aldehyde dehydrogenase-expressing progenitor cells promote recovery from acute ischemic injury. Stem Cells. 2012 Oct;30(10):2248-60. doi: 10.1002/stem.1206. PMID 22899443
- [Result] Hess DA, Meyerrose TE, Wirthlin L, Craft TP, Herrbrich PE, Creer MH, Nolta JA. Functional characterization of highly purified human hematopoietic repopulating cells isolated according to aldehyde dehydrogenase activity. Blood. 2004 Sep 15;104(6):1648-55. doi: 10.1182/blood-2004-02-0448. Epub 2004 Jun 3. PMID 15178579
- [Result] Fallon P, Gentry T, Balber AE, Boulware D, Janssen WE, Smilee R, Storms RW, Smith C. Mobilized peripheral blood SSCloALDHbr cells have the phenotypic and functional properties of primitive haematopoietic cells and their number correlates with engraftment following autologous transplantation. Br J Haematol. 2003 Jul;122(1):99-108. doi: 10.1046/j.1365-2141.2003.04357.x. PMID 12823351
- [Result] Hess DA, Wirthlin L, Craft TP, Herrbrich PE, Hohm SA, Lahey R, Eades WC, Creer MH, Nolta JA. Selection based on CD133 and high aldehyde dehydrogenase activity isolates long-term reconstituting human hematopoietic stem cells. Blood. 2006 Mar 1;107(5):2162-9. doi: 10.1182/blood-2005-06-2284. Epub 2005 Nov 3. PMID 16269619
- [Result] Putman DM, Cooper TT, Sherman SE, Seneviratne AK, Hewitt M, Bell GI, Hess DA. Expansion of Umbilical Cord Blood Aldehyde Dehydrogenase Expressing Cells Generates Myeloid Progenitor Cells that Stimulate Limb Revascularization. Stem Cells Transl Med. 2017 Jul;6(7):1607-1619. doi: 10.1002/sctm.16-0472. Epub 2017 Jun 15. PMID 28618138
- [Result] Perin EC, Murphy MP, March KL, Bolli R, Loughran J, Yang PC, Leeper NJ, Dalman RL, Alexander J, Henry TD, Traverse JH, Pepine CJ, Anderson RD, Berceli S, Willerson JT, Muthupillai R, Gahremanpour A, Raveendran G, Velasquez O, Hare JM, Hernandez Schulman I, Kasi VS, Hiatt WR, Ambale-Venkatesh B, Lima JA, Taylor DA, Resende M, Gee AP, Durett AG, Bloom J, Richman S, G'Sell P, Williams S, Khan F, Gyang Ross E, Santoso MR, Goldman J, Leach D, Handberg E, Cheong B, Piece N, DiFede D, Bruhn-Ding B, Caldwell E, Bettencourt J, Lai D, Piller L, Simpson L, Cohen M, Sayre SL, Vojvodic RW, Moye L, Ebert RF, Simari RD, Hirsch AT; Cardiovascular Cell Therapy Research Network (CCTRN). Evaluation of Cell Therapy on Exercise Performance and Limb Perfusion in Peripheral Artery Disease: The CCTRN PACE Trial (Patients With Intermittent Claudication Injected With ALDH Bright Cells). Circulation. 2017 Apr 11;135(15):1417-1428. doi: 10.1161/CIRCULATIONAHA.116.025707. Epub 2017 Feb 16. PMID 28209728
- [Result] Terenzi DC, Al-Omran M, Quan A, Teoh H, Verma S, Hess DA. Circulating Pro-Vascular Progenitor Cell Depletion During Type 2 Diabetes: Translational Insights Into the Prevention of Ischemic Complications in Diabetes. JACC Basic Transl Sci. 2018 Nov 5;4(1):98-112. doi: 10.1016/j.jacbts.2018.10.005. eCollection 2019 Feb. PMID 30847424
- [Result] Hess DA, Terenzi DC, Trac JZ, Quan A, Mason T, Al-Omran M, Bhatt DL, Dhingra N, Rotstein OD, Leiter LA, Zinman B, Sabongui S, Yan AT, Teoh H, Mazer CD, Connelly KA, Verma S. SGLT2 Inhibition with Empagliflozin Increases Circulating Provascular Progenitor Cells in People with Type 2 Diabetes Mellitus. Cell Metab. 2019 Oct 1;30(4):609-613. doi: 10.1016/j.cmet.2019.08.015. Epub 2019 Aug 30. PMID 31477497
- [Result] Hess DA, Trac JZ, Glazer SA, Terenzi DC, Quan A, Teoh H, Al-Omran M, Bhatt DL, Mazer CD, Rotstein OD, Verma S. Vascular Risk Reduction in Obesity through Reduced Granulocyte Burden and Improved Angiogenic Monocyte Content following Bariatric Surgery. Cell Rep Med. 2020 May 19;1(2):100018. doi: 10.1016/j.xcrm.2020.100018. eCollection 2020 May 19. PMID 33205058
- See also: IDF Diabetes atlas, 10th ed. — http://www.ncbi.nlm.nih.gov/books/NBK581934/